CLINICAL TRIAL: NCT04142905
Title: Is Asthma in Subjects With Obstructive Sleep Apnoea (OSA) Due to Dysanapsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Julie Dawson (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 269072
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Asthma; Obstructive Sleep Apnoea (OSA); Dysanapis
MeSH Terms: conditions — Asthma; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients With Asthma: Subjects with sleep disordered breathing with asthma
- Patients Without Asthma: Subjects with sleep disordered breathing without asthma

SUMMARY:
Intention to review patient letters from sleep clinic to see if their lung function fit in with Dysynapsis in wheezing patients or if it is true asthma

DETAILED DESCRIPTION:
There is no evidence that the World Wide prevalence of asthma is declining. There is some evidence that this Western disease may give the appearance of declining prevalence due to improved healthcare. However evidence from the Office of National Statistics suggests that the mortality rate for asthma may be increasing year on since 2007 until 2017. The true burden of asthma in the United Kingdom is difficult to ascertain.

Obesity has effects on lung function which lead to low functional residual capacity and low end reserve volume. This leads to rapid shallow breaths near to the airway closing pressure and lung closing volume as illustrated in this review. This suggests that obesity itself may be a source of breathlessness.

High Body Mass Index (BMI) has been shown to be associated with asthma. It was also associated with wheeze that is not asthma. This finding suggests that obesity in itself may be linked to wheeze which is not asthma. It has been shown in children that sleep disordered breathing is associated with asthma as well as wheeze. Obese children are known to display dysanapsis (airway cross sectional area is small for the size of the lung) whether associated with or without asthma, however if associated with asthma, the severity of asthma can be worse.

AIM: To investigate if asthma is truly associated with Sleep disordered breathing in adult subjects. To investigate if there is an association of wheeze with dysanapsis in patients with sleep disordered breathing

NULL HYPOTHESIS: There is no difference between subjects who have sleep disordered breathing with asthma and those subjects who have sleep disordered breathing without asthma, with respect to lung function parameters.

Methods

Initially the investigators' aim is to interrogate clinical records and look at lung function testing in subjects with and without asthma who attend the sleep disordered breathing clinic. The investigators intend to investigate 100 with asthma in the sleep clinic and 100 without asthma in the sleep clinic. The Investigators will also look at eosinophil results of those with asthma compared to those without asthma and any markers of atopy.

The investigators will use Statistical Package for the Social Sciences (SPSS) to undertake simple frequency analysis and cross tabs as well as odds ratio from binary logistic regression.

References - Refer to References Section

Appendix 1

Data Collection Sheet for those with confirmed diagnosis of Obstructive sleep apnoea

Name and Date of Birth and details

Age

Weight ______Height___________Body Mass Index _________Gender at birth ___Male____Female___ Asthma diagnosis made by General Practitioner or Respiratory physician or no diagnosis of asthma (circle correct)

DATE of Test ___/___/___FEV1_______FEV1%_______

FVC_________FVC%__________

DATE of Test ___/___/___FEV1_______FEV1%_______

FVC_________FVC%__________

Dysanapsis FEV1/FVC <0.8 Yes/No FEV1/FVC <0.7 Yes/No (circle correct)

AHI/hr 5-15 16-29 >30 (circle correct)

Eosinophil count MAX in past 12 months________x109/L MAX ever ______ x109/L

DATE________

RAST test positive for which antigens

Smoking history start age________________ Pack years________________

ELIGIBILITY:
Inclusion Criteria:

* Any subject in Obstructive Sleep Apnea clinic.

Exclusion Criteria:

* Only exclusion criteria is if they have no recorded lung function in their notes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients attending the Obstructive Sleep Apnea Clinic at Norfolk & Norwich University Hospital NHS Foundation Trust
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Defined dysynapsis in patients with asthma and obstructive sleep apnoea (OSA) | 6 years
  The investigator will refer to the Sleep Disordered Breathing Clinic records to investigate the prevalence of dysanapsis in patients with Sleep disordered breathing, in patients with asthma compared to those without asthma.

SECONDARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 6 years
  The investigator will refer to the Sleep Disordered Breathing Clinic records to compare measures of Apnea-Hypopnea Index (AHI) in patients with and without asthma.
Eosinophil count | 6 years
  The investigator will refer to the Sleep Disordered Breathing Clinic records to compare Eosinophil count in patients with and without asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, United Kingdom

REFERENCES:
- [Background] Anandan C, Nurmatov U, van Schayck OC, Sheikh A. Is the prevalence of asthma declining? Systematic review of epidemiological studies. Allergy. 2010 Feb;65(2):152-67. doi: 10.1111/j.1398-9995.2009.02244.x. Epub 2009 Nov 12. PMID 19912154
- [Background] Mukherjee M, Gupta R, Farr A, Heaven M, Stoddart A, Nwaru BI, Fitzsimmons D, Chamberlain G, Bandyopadhyay A, Fischbacher C, Dibben C, Shields M, Phillips C, Strachan D, Davies G, McKinstry B, Sheikh A; Burden and True Cost of Asthma in the UK Research Team. Estimating the incidence, prevalence and true cost of asthma in the UK: secondary analysis of national stand-alone and linked databases in England, Northern Ireland, Scotland and Wales-a study protocol. BMJ Open. 2014 Nov 4;4(11):e006647. doi: 10.1136/bmjopen-2014-006647. PMID 25371419
- [Background] Jones RL, Nzekwu MM. The effects of body mass index on lung volumes. Chest. 2006 Sep;130(3):827-33. doi: 10.1378/chest.130.3.827. PMID 16963682
- [Background] Beuther DA, Weiss ST, Sutherland ER. Obesity and asthma. Am J Respir Crit Care Med. 2006 Jul 15;174(2):112-9. doi: 10.1164/rccm.200602-231PP. Epub 2006 Apr 20. PMID 16627866
- [Background] von Mutius E, Schwartz J, Neas LM, Dockery D, Weiss ST. Relation of body mass index to asthma and atopy in children: the National Health and Nutrition Examination Study III. Thorax. 2001 Nov;56(11):835-8. doi: 10.1136/thorax.56.11.835. PMID 11641506
- [Background] Colak Y, Afzal S, Lange P, Nordestgaard BG. Obese individuals experience wheezing without asthma but not asthma without wheezing: a Mendelian randomisation study of 85,437 adults from the Copenhagen General Population Study. Thorax. 2016 Mar;71(3):247-54. doi: 10.1136/thoraxjnl-2015-207379. Epub 2015 Oct 26. PMID 26504195
- [Background] Sulit LG, Storfer-Isser A, Rosen CL, Kirchner HL, Redline S. Associations of obesity, sleep-disordered breathing, and wheezing in children. Am J Respir Crit Care Med. 2005 Mar 15;171(6):659-64. doi: 10.1164/rccm.200403-398OC. Epub 2004 Dec 10. PMID 15591475
- [Background] Forno E, Weiner DJ, Mullen J, Sawicki G, Kurland G, Han YY, Cloutier MM, Canino G, Weiss ST, Litonjua AA, Celedon JC. Obesity and Airway Dysanapsis in Children with and without Asthma. Am J Respir Crit Care Med. 2017 Feb 1;195(3):314-323. doi: 10.1164/rccm.201605-1039OC. PMID 27552676